CLINICAL TRIAL: NCT03415685
Title: Evaluation of the Lutronic PicoPlus for the Treatment of Dematological Conditions Such as Unwanted Tattoos and Benign Pigmented Lesions
Brief Title: Lutronic PicoPlus Exploratory Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped due to pivot in company clinical strategy.
Sponsor: CynosureLutronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L16004
Record Dates: First submitted 2018-01-08; First posted 2018-01-30 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Tattoo; Pigmentation; Melasma; Benign Pigmented Lesion
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to one of two treatments group depending on the dermatologic condition to be treated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A: PicoPlus for unwanted tattoos. (Active Comparator): Subjects receiving PicoPlus laser system treatment for unwanted tattoos.
  Interventions: Device: PicoPlus laser system
- Group B: PicoPlus for other dermatological conditions (Active Comparator): Subjects receiving PicoPlus laser system treatment for unwanted benign pigmented lesions, melasma or other dermatological conditions such as skin rejuvenation.
  Interventions: Device: PicoPlus laser system

INTERVENTIONS:
Device: PicoPlus laser system — Laser treatment using specific pulse durations and wavelengths for selective pigment photothermolysis.

SUMMARY:
This study will evaluate the use of the Lutronic PicoPlus for treatment of dermatological conditions such as unwanted tattoos and benign pigmented lesions.

DETAILED DESCRIPTION:
This pilot clinical trial will evaluate the capability of the Lutronic PicoPlus technology to remove unwanted tattoos and benign pigmented lesions. This trial is designed as a multi-center exploratory, open-label clinical trial comparing each subject's condition before and after treatment. Subjects meeting all entrance criteria will be assigned to Group A for treatment of unwanted tattoos and Group B for treatment of unwanted benign pigmented lesions, melasma, or other skin conditions such as skin rejuvenation. Subjects in each treatment group will receive a series of treatments, e.g., 2-5, and will be asked to complete 1 and 3 month follow-up visit(s) following each treatment to assess treatment efficacy and safety. At investigators' discretion, additional follow-up visits, e.g., at 6 months following treatment, may take place to observe the time course of reactions after treatment and/or assess efficacy. Outcome measures include clinician grading and subject satisfaction post-treatment. Pre-treatment study photos will be obtained at baseline; post-treatment study photos will be obtained at each post-treatment follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Adults between age 18 and 60 years old
* Group A: Fitzpatrick skin type I - VI for unwanted tattoos and Group B: Fitzpatrick Skin Types I - IV for benign pigmented lesions and other conditions
* Unwanted tattoo that contains single or multi-color ink, and

  * Wiling to cover tattoos with a bandage or clothing; and/or have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treated area starting 2 to 4 weeks before the treatment
* Ability to read, understand, and sign the Informed Consent Form
* Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated
* Willing and able to comply with all study participation requirements including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study

Exclusion Criteria:

* If receiving treatment for unwanted tattoo: double tattoos (tattoo over tattoo), history of allergic reactions to pigments following tattooing, local anesthetics or topical antibiotics
* If receiving treatment for benign pigmented lesions including melasma: history of use of a lightening medication (hydroquinone, tranexamic acid), isotretinoid (or retinoid), or light-sensitive medication in the last 6 months
* Known cardiovascular disease or cardiac surgery that in the opinion of the investigator would interfere with study treatments
* Previous interventions or treatment with another device in the target area within 6 months of enrollment or during the study
* Pregnant or lactating or planning pregnancy before end of study
* Presence of an active systemic, local skin disease, medication or condition that may affect wound healing or interfere with participation or treatment to the active area.
* Active or recurrent cancer of current chemotherapy or radiation therapy
* History of seizure disorders due to light
* History of vitiligo, eczema, or psoriasis
* History of connective tissue disease, such as systemic lupus erythematosus or scleroderma
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation
* History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
* History of seizure disorders due to light.
* Suffering from coagulation disorders or taking prescription anticoagulation medications
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing Any use of medication that is known to increase sensitivity to light according to Investigator's discretion
* Excessive or recent significant tan in areas to be treated or unable/unlikely to refrain from tanning during the study
* Current smoker or history of smoking within 3 months of study participation
* Systemic use of corticosteroid or isotretinoin within 6 months of study participation
* Anytime in life, having have used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus
* Any physical or mental condition including alcohol or drug abuse that in the opinion of the investigator could interfere with subject's suitability for inclusion in study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari Larson, MBA, Study Director — Sponsor GmbH
Locations (4):
- United States (4):
  - Zena Medical, Newport Beach, California
  - Metro Dermatology, Elmhurst, New York
  - Laser and Skin Surgery Center of New York, New York, New York
  - Dermatology, Laser, and Vein Specialists of the Carolinas, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were assigned a group depending on the condition that was to be treated as part of their participation in the study.
Groups:
- Group A: PicoPlus for Unwanted Tattoos.: Subjects receiving PicoPlus laser system treatment for unwanted tattoos. Subjects can receive up to 8 treatments with a standard interval of 6-8 weeks between treatments.
  PicoPlus laser system: Laser treatment using specific pulse durations and wavelengths for selective pigment photothermolysis.
- Group B: PicoPlus for Other Dermatological Conditions: Subjects receiving PicoPlus laser system treatment for unwanted benign pigmented lesions, melasma or other dermatological conditions such as skin rejuvenation.
  Subjects can receive up to 8 treatments with a standard interval of 3-5 weeks between treatments.
  PicoPlus laser system: Laser treatment using specific pulse durations and wavelengths for selective pigment photothermolysis.
Period: Overall Study
Arm/Group | Group A: PicoPlus for Unwanted Tattoos. | Group B: PicoPlus for Other Dermatological Conditions
Started | 11 | 28
Completed | 11 | 9
Not Completed | 0 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: PicoPlus for Unwanted Tattoos. | Group B: PicoPlus for Other Dermatological Conditions | Total
Number analyzed (Participants) | 11 | 28 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (6.9) | 43.6 (15.4) | 38.7 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 28 | 36
  Male | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 11 | 15 | 26
  Unknown or Not Reported | 0 | 9 | 9

OUTCOME MEASURES:

1. Primary Outcome: Investigator's Global Assessment of Improvement
Description: Overall aesthetic improvement based on completion of the Physician's Global Assessment of Improvement Scale. Physician evaluators will review study photos post-final treatment, and rate the degree of tattoo clearing or reduction in benign pigmentation observed in the subject's treated area using the following definitions:
  3 = Very significant or complete clearing (75-100%)
  2 = Significant clearing (50-74%)
  1 = Moderate clearing (25-49%)
  0 = Mild or no clearing (0-24%)
Time Frame: Up to 6 Months following final study treatment
Population: # of subjects who returned for FU assessment prior to study termination
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: PicoPlus for Unwanted Tattoos. | Group B: PicoPlus for Other Dermatological Conditions
Number analyzed (Participants) | 6 | 8
Participants
  3 = Very significant or complete clearing (75-100%) | 1 | 6
  2 = Significant clearing (50-74%) | 2 | 0
  1 = Moderate clearing (25-49%) | 3 | 2
  0 = Mild or no clearing (0-24%) | 0 | 0

2. Secondary Outcome: Subject's Global Assessment of Improvement
Description: Overall aesthetic improvement based on completion of the Subject's Global Assessment of Improvement Scale. Subjects will be asked review study photos post-final treatment, and rate the degree of tattoo clearing or reduction in benign pigmentation observed in the subject's treated area using the following definitions:
  3 = Very significant or complete clearing (75-100%)
  2 = Significant clearing (50-74%)
  1 = Moderate clearing (25-49%)
  0 = Mild or no clearing (0-24%)
Time Frame: 1 month, 3 Months, 6 Months (Group A Only) post final treatment
Population: A subset of subjects (6 in Group A, 9 in Group B) returned for a 1-month follow-up prior to termination of the study with results reported in the corresponding table.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: PicoPlus for Unwanted Tattoos. | Group B: PicoPlus for Other Dermatological Conditions
Number analyzed (Participants) | 6 | 9
Participants
  3 = Very significant or complete clearing (75-100%) | 0 | 6
  2 = Significant clearing (50-74%) | 3 | 3
  1 = Moderate clearing (25-49%) | 3 | 0
  0 = Mild or no clearing (0-24%) | 0 | 0

3. Secondary Outcome: Subject Satisfaction
Description: Following the final study treatment, subjects will be asked to rate their level of satisfaction with the laser treatment outcome and the overall laser treatment procedure, using the Subject Satisfaction Assessment Scale and the following definitions:
  2 = Extremely Satisfied
  1 = Satisfied
  0 = Neutral
  (-1) = Unsatisfied
  (-2) = Extremely Unsatisfied
Time Frame: 1 month, 3 Months, 6 Months (Group A Only) post final treatment
Population: Data cannot be reported as satisfaction data was not collected at the time of patient visits.
Arm/Group | Group A: PicoPlus for Unwanted Tattoos. | Group B: PicoPlus for Other Dermatological Conditions
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Blinded Reviewer's Global Assessment of Improvement
Description: Three blinded experienced, non-treating clinicians will independently evaluate pre- and post-treatment photos of each subject, presented randomly. Each reviewer will be asked to determine the temporal order (before and after) of each photo pair, and then rate the degree of tattoo clearing or reduction in benign pigmentation in the post-treatment photo using the following scale:
  3 = Very significant or complete clearing (75-100%)
  2 = Significant clearing (50-74%)
  1 = Moderate clearing (25-49%)
  0 = Mild or no clearing (0-24%)
Time Frame: 3-month (Group B), 6 months (Group A) Post Final treatment
Population: Due to study termination a blinded review was not completed for the subject images in the study and thus there is no data to report.
Arm/Group | Group A: PicoPlus for Unwanted Tattoos. | Group B: PicoPlus for Other Dermatological Conditions
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Melasma Area Severity Index (MASI)
Description: Three blinded experienced, non-treating clinicians will independently evaluate pre- and post-treatment photos of each subject, presented randomly, using the MASI. Each of four regions (forehead, right malar region, left malar region and chin) will be assessed based on three variables: percentage of the total area involved (A), darkness (D), and homogeneity (H).
Time Frame: 3 Months (Group B), 6 Months (Group A) post final treatment
Population: MASI scoring was not completed for participants in the study as the study was terminated and Blinded Reviewers did not evaluate the photos.
Arm/Group | Group A: PicoPlus for Unwanted Tattoos. | Group B: PicoPlus for Other Dermatological Conditions
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 6 months post final treatment.
Arm/Group | Group A: PicoPlus for Unwanted Tattoos. | Group B: PicoPlus for Other Dermatological Conditions
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/28
Other Adverse Events (participants affected / at risk) | 2/11 | 11/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: PicoPlus for Unwanted Tattoos. (N=11) | Group B: PicoPlus for Other Dermatological Conditions (N=28)
Darkening of Lesions (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (8)
Blisters/Scabs/Crusting (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Bruising/Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Edema (Skin and subcutaneous tissue disorders) | 1 (3) | 7 (13)
Erythema (Skin and subcutaneous tissue disorders) | 2 (4) | 10 (23)
Bleeding of Ink (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Treatment Discomfort (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dryness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Heat Sensation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Hypo/Hyper-Pigmentation (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3)
Itching/Pruritis (Skin and subcutaneous tissue disorders) | 2 (6) | 5 (6)
Skin Bumps (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Roughness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scabbing/Peeling (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Tightness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Welting/Raised Area of Edema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of the study led to reduced endpoint evaluation and consistent timing for all the endpoints which were analyzed. It also means that full treatment regimen to fully observe the treatment effectiveness and safety could not be fully completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT03415685/Prot_000.pdf